CLINICAL TRIAL: NCT06865859
Title: Single-cell Landscape of Immunological Responses in Patients with Hepatitis B Virus-related Acute-on-chronic Liver Failure
Brief Title: Single Cell Landscape of HBV-related Acute-on-chronic Liver Failure Patients
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202310-036
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-04

CONDITIONS: HBV Related Acute-on-chronic Liver Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood and liver tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Chronic Hepatitis B
- HBV related liver cirrhosis
- HBV related acute-on-chronic hepatic dysfunction
- HBV related acute-on-chronic liver failure

SUMMARY:
This study aimed to profile the peripheral blood immune cells of patients with HBV related acute-on-chronic liver failure using single-cell RNA sequencing to reveal the immunopathological mechanisms of HBV related acute-on-chronic liver failure.

DETAILED DESCRIPTION:
Acute-on-chronic liver failure (ACLF) is a complex clinical syndrome characterized by acute deterioration of liver function in patients with chronic liver disease, exhibiting liver and extrahepatic organ failure and a high short-term mortality. Immune imbalance plays an important role in the progression of HBV-related ACLF. Further investigation of the immune cell characteristics of HBV-related ACLF is helpful to understand its pathogenesis, and may provide reference for the effective therapeutic agent. Single-cell RNA sequencing (scRNA-seq) is the quantitative analysis of transcription at the single-cell level, which could provide systematic analyses of transcriptomic profiles, infer cell-cell interactions. This study will combine single cell transcriptomics and molecular biological experiment to elucidate the immunopathological cell states associated with HBV-related chronic liver disease vs. ACLF.

ELIGIBILITY:
Inclusion Criteria:

Acute liver failure is a well-defned medical emergency which is defned as a severe liver injury, leading to coagulation abnormality usually with an INR ≥ 1.5, and any degree of mental alteration (encephalopathy) in a patient without pre-existing liver disease and with an illness of up to 4 weeks duration

Exclusion Criteria:

* Associated with other types of hepatitis virus infection or HIV infection, alcoholic liver disease, autoimmune liver disease, drug-induced liver injury; ② Suffering from primary liver cancer or severe heart, digestive, lung, kidney, neurological and psychiatric diseases; ③ Patients with incomplete data and patients unable to participate in the experiment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is patients with chronic hepatitis B，HBV related liver cirrhosis，HBV related acute-on-chronic hepatic dysfunction and HBV related acute-on-chronic liver failure
Sampling Method: Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Mortality | 28 days, 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No